CLINICAL TRIAL: NCT06397183
Title: Comparison Of Mulligan Stretch With Traction Technique And Post Isometric Relaxation On Hamstring Flexibility In Athletes
Brief Title: Mulligan Stretch With Traction Versus Post Isometric Relaxtion on Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/21/0419
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hamstring Flexibility
Keywords: Hamstring Flexibility; Sports Injury; Muscle Energy Technique; Post Isometric Relaxation
MeSH Terms: conditions — Athletic Injuries | interventions — Traction; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Strech with Traction Group (Experimental)
  Interventions: Other: Mulligan Strech with Traction (TSLR) Technique
- Post-Isometric Relaxation Group (Experimental)
  Interventions: Other: Post-Isometric Relaxation Technique

INTERVENTIONS:
Other: Mulligan Strech with Traction (TSLR) Technique — The Mulligan traction straight leg raise (TSLR) technique is a mobilization technique that can increase hamstring flexibility and range of motion.
  Arms: Mulligan Strech with Traction Group
Other: Post-Isometric Relaxation Technique — Post-Isometric Relaxation Technique is a Muscle Energy Technique which increases hamstring flexibility and range of motion.
  Arms: Post-Isometric Relaxation Group

SUMMARY:
The design of my study will be Randomized Control Trial (RCT) study. And the sampling technique will be non-probability convenience sampling. A sample of 32 (16 in each group) has been selected using 10% level of significance and 80% power of test.

Three groups will be made each containing 16 participants with inclusion criteria met. Group A will be given control group treatment with Muscle Energy Technique applied over the period of 4 weeks. Group B will be given control group treatment with Mulligan Stretch with Traction Technique applied over the period of 4 weeks.

Total 3 recordings of Hip Flexion ROMs shall be taken with manual goniometry as follows initial/first day, 3rd week, final week/last treatment. A sum of 8 treatments shall be given to the intervention group over the period of 4 weeks, 2 treatments per week.

DETAILED DESCRIPTION:
INTRODUCTION:

Mobility in human gait depends on flexibility of hamstring muscles. Hamstring muscles function is hip extension and knee flexion. In most of the population, tightness or shortening of hamstring muscles occur which limits hip flexion. To measure hamstring muscles flexibility simple passive SLR is performed and range is recorded by manual goniometer. To increase SLR, several techniques are used: MET's and TSLR. Effectiveness of these techniques depend on muscle flexibility.

OBJECTIVE:

The purpose of this study is to compare the effectiveness of mulligan stretch with traction technique and muscle energy technique to increase the SLR in athletes with hamstring tightness.

METHOD:

The data will be collected from Athletes in sports clubs, gyms, and sports fields of Lahore. The study will be completed in a period of six months after the approval of synopsis. The design of my study will be Randomized Control Trial (RCT) study. And the sampling technique will be non-probability convenience sampling. A sample of 32 (16 in each group) has been selected using 10% level of significance and 80% power of test.

Three groups will be made each containing 16 participants with inclusion criteria met. Group A will be given control group treatment with Muscle Energy Technique applied over the period of 4 weeks. Group B will be given control group treatment with Mulligan Stretch with Traction Technique applied over the period of 4 weeks.

Total 3 recordings of Hip Flexion ROMs shall be taken with manual goniometry as follows initial/first day, 3rd week, final week/last treatment. A sum of 8 treatments shall be given to the intervention group over the period of 4 weeks, 2 treatments per week.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Negative Spring test
* Asymptomatic
* SLR < 80⸰

Exclusion Criteria:

* Positive LBP
* Lumbar Straightening
* SI Joint Dysfunction
* History of hamstring injury
* Current musculoskeletal pain in hip region
* Any other comorbidity limiting joint ROM

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Hip Flexion Range of Motion | Baseline, 3rd week and 6th week.
  Hip Flexion ROM will be measured using SLR technique with manual goniometry.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Shapes Executive Gym Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No